CLINICAL TRIAL: NCT02018939
Title: Multiple-dose Pharmacokinetics of Doripenem During Continuous Venovenous Hemodiafiltration and Molecular Adsorbent Recirculating System in ICU Patients and During Hemodialysis in Longterm Hemodialysis Patients.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Florian Thalhammer, a.o.Univ.-Prof. Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DORIPENEM IN CVVH, MARS AND HD
Record Dates: First submitted 2013-10-16; First posted 2013-12-23 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Infections During Organ Replacement Therapy
Keywords: pharmacokinetics, doripenem, renal replacement therapy, MARS, organ replacement therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Pharmacokinetic profiling in Hemodialysis (Experimental): Patients with chronic intermittent hemodialysis receiving doripenem therapy are included in this arm. Pharmacokinetic samples are drawn.
  Interventions: Other: Pharmacokinetic profiling
- Pharmacokinetic profiling in CVVH (Experimental): Patients receiving continuous venovenous renal replacement therapy in an ICU setting receiving doripenem therapy are included in this arm. Pharmacokinetic samples are drawn.
  Interventions: Other: Pharmacokinetic profiling
- Pharmacokinetic profiling in MARS (Experimental): Patients receiving liver replacement therapy (MARS) in an ICU setting receiving doripenem therapy are included in this arm. Pharmacokinetic samples are drawn.
  Interventions: Other: Pharmacokinetic profiling

INTERVENTIONS:
Other: Pharmacokinetic profiling — Pharmacokinetic samples are taken from each Patient receiving Doripenem in each arm. No other interventions are performed during this trial. Doripenem is not administered due to the trial.

SUMMARY:
The study is conducted to investigate the pharmacokinetics of Doripenem during CVVHDF (Continuous venovenous hemodiafiltration), MARS (Molecular Adsorbent Recirculating System) and intermittent hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Suspected or proven bacterial infection requiring parenteral antibiotic therapy.
* Organ replacement therapy (MARS, CVVHDF or HD)

Exclusion Criteria:

* Known hypersensitivity to doripenem or other carbapenems, or severe hypersensitivity (anaphylactic reaction) to beta-lactam antibacterial agents.
* An expected survival of less than two days.
* Known pregnancy
* Coadministration of valproic acid or probenecid, which cannot be discontinued for the duration of the study
* Doripenem as monotherapy for resistent species or fungal infections.
* Other reasons opposing the study participation on the discretion of the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Influence of organ replacement therapy on area under curve of doripenem serum concentration | day 15
  Pharmacokinetic samples are drawn from each patient during the trial. Analysis by HPLC will be conducted after the end of the trial.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Derived] Vossen MG, Ehmann L, Pferschy S, Maier-Salamon A, Haidinger M, Weiser C, Wenisch JM, Saria K, Kajahn C, Jilch S, Lemmerer R, Becede M, Zeitlinger M, Kloft C, Jager W, Thalhammer F. Elimination of Doripenem during Dialysis and Pharmacokinetic Evaluation of Posthemodialysis Dosing for Patients Undergoing Intermittent Renal Replacement Therapy. Antimicrob Agents Chemother. 2018 Apr 26;62(5):e02430-17. doi: 10.1128/AAC.02430-17. Print 2018 May. PMID 29530855
- [Derived] Vossen MG, Wenisch JM, Maier-Salamon A, Fritsch A, Saria K, Zuba C, Jilch S, Lemmerer R, Unger M, Jaehde U, Jager W, Thalhammer F. Doripenem Treatment during Continuous Renal Replacement Therapy. Antimicrob Agents Chemother. 2015 Dec 28;60(3):1687-94. doi: 10.1128/AAC.01801-15. PMID 26711775